CLINICAL TRIAL: NCT02843061
Title: Combination of Rituximab and NK Immunotherapy for B Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: Shenzhen Hank Bioengineering Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NK-Rituximab
Record Dates: First submitted 2016-07-21; First posted 2016-07-25 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-07

CONDITIONS: B-cell Lymphoma Recurrent
Keywords: B lymphoma; Rituximab; NK immunotherapy
MeSH Terms: interventions — Rituximab

ARMS (2):
- Rituximab and NK immunotherapy (Experimental): In this group, the patients will receive regular Rituximab treatment accompanied with multiple NK immunotherapy. The check indexes are CT scan and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).
  Interventions: Drug: Rituximab; Biological: NK immunotherapy
- Rituximab (Active Comparator): In this group, the patients will receive regular Rituximab to decrease tumor burden. The check indexes are CT scan and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab
  Other Names: IDEC-C2B8 or Rituxan
Biological: NK immunotherapy — Each time 10 billion cells, 4 times in all,i.v.
  Other Names: natural killer cell
  Arms: Rituximab and NK immunotherapy

SUMMARY:
The aim of this study is the safety and efficacy of Rituximab plus NK immunotherapy to recurrent B lymphoma.

DETAILED DESCRIPTION:
By enrolling patients with B lymphoma adapted to enrolled criteria, this study will document for the first time the safety and the short and long term efficacy of the combined therapy using Rituximab and natural killer (NK) cells.

The safety will be evaluated by statistics of adverse reactions. The efficacy will be evaluated according to local relief degree, progress free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* All standard therapies have failed according to NCCN guidelines or the patient refuses standard therapies after cancer recurrence
* Body tumor 1-6, the maximum tumor length < 5 cm
* KPS ≥ 70, lifespan > 6 months
* Platelet count ≥ 80×109/L，white blood cell count ≥ 3×109/L, neutrophil count ≥ 2×109/L, hemoglobin ≥ 80 g/L

Exclusion Criteria:

* Patients with cardiac pacemaker
* Patients with brain metastasis
* Patients with grade 3 hypertension or diabetic complication, severe cardiac and pulmonary dysfunction

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Relief degree evaluated by the RECIST | 3 months
  It will be evaluated by the Response Evaluation Criteria in Solid Tumors (RECIST)

SECONDARY OUTCOMES:
Progress free survival (PFS) | 1 year
Overall survival (OS) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jibing Chen, MD, PhD, Principal Investigator — Fuda Cancer Hospital, Guangzhou
Locations (1):
- Cancer Institute in Fuda cancer hospital, Guangzhou, Guangdong, China